CLINICAL TRIAL: NCT00020007
Title: A Phase I Study of Isolated Lung Perfusion With Paclitaxel and Moderate Hyperthermia in Patients With Unresectable Pulmonary Malignancies
Brief Title: Paclitaxel and Hyperthermic Perfusion in Treating Patients With Lung Cancer or Lung Metastases That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067490; NCI-00-C-0019; NCT00001939 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2006-01

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: recurrent non-small cell lung cancer; limited stage small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; lung metastases; bronchoalveolar cell lung cancer; pulmonary carcinoid tumor
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Paclitaxel; Diathermy

INTERVENTIONS:
Drug: isolated perfusion
Drug: paclitaxel
Procedure: hyperthermia treatment

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Heating paclitaxel to several degrees above body temperature and infusing it to the affected area around the tumor may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of paclitaxel given by hyperthermic perfusion in treating patients with lung cancer or lung metastases that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and phase II dose of paclitaxel administered via hyperthermic retrograde isolated lung perfusion in patients with unresectable pulmonary malignancies.
* Determine the nature of the toxic effects of this regimen in this patient population.
* Evaluate the pharmacokinetic profile of this regimen in these patients.
* Determine the relationship between pharmacodynamic parameters and toxic effects of this regimen in these patients.

OUTLINE: This is a dose-escalation study of paclitaxel.

Patients undergo posterolateral thoracotomy or median sternotomy. Patients receive paclitaxel over 90 minutes administered via hyperthermic retrograde isolated lung perfusion. The entire surgery lasts approximately 4 hours.

Cohorts of 3-6 patients receive escalating doses of paclitaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 1 and 2 months. Patients with responding disease continue to be followed every 3 months.

PROJECTED ACCRUAL: A maximum of 31 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed unresectable primary lung cancer or pulmonary metastases that are unresectable on the basis of technical considerations or are sufficiently numerous that recurrent, potentially inoperable disease is highly probable

  * Bilateral metastases allowed
  * Unresectable bronchoalveolar carcinomas allowed
  * Previously treated primary lung cancer allowed
* Disease outside confines of thorax allowed, provided bulk of disease in the chest is clearly the greatest threat to survival and/or extrathoracic disease is controlled
* No potentially treatable pulmonary metastases from lymphomas or germ cell tumors
* No biopsy proven interstitial fibrosis, radiation induced pneumonitis, or evidence of significant pulmonary hypertension by history, radiologic, echocardiographic, or catheterization studies
* No active intracranial or leptomeningeal metastases

  * Prior resection or radiotherapy for intracranial metastases allowed if the following criteria are met:

    * No active disease on 2 MRIs done one month apart
    * No requirement for anticonvulsant medications or steroids
* Adequate pulmonary reserve to tolerate pneumonectomy:

  * Oxygen consumption greater than 50% predicted AND
  * FEV1 and DLCO greater than 80% predicted OR
  * FEV1 or DLCO less than 80% predicted allowed if postoperative FEV1 and DLCO is at least 40% predicted on the basis of split function V/Q scan
* Prior radiotherapy to chest allowed provided 6 months have elapsed since completion of treatment and no history of, nor current evidence of, interstitial lung disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* More than 3 months

Hematopoietic:

* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10 g/dL
* WBC greater than 3,500/mm^3

Hepatic:

* PT/PTT normal
* Bilirubin less than 1.5 times upper limit of normal (ULN)
* AST/ALT less than 1.5 times ULN

Renal:

* Creatinine less than 1.6 mg/dL

Cardiovascular:

* Fixed defects on thallium scanning with ejection fraction greater than 40% allowed
* Reversible or ischemic defects allowed only after cardiology clearance

Pulmonary:

* See Disease Characteristics
* Resting oxygen saturation greater than 90%
* pCO_2 less than 45 mmHg by arterial blood gas

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infections
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* More than 30 days since prior biologic therapy for this malignancy

Chemotherapy:

* More than 30 days since prior chemotherapy for this malignancy
* Prior paclitaxel allowed
* No prior bleomycin, nitrosoureas, or busulfan

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics
* Prior thoracic surgery allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12

CONTACTS AND LOCATIONS:
Overall Officials: David S. Schrump, MD, Study Chair — NCI - Surgery Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland